CLINICAL TRIAL: NCT04651361
Title: Efficacy of Preoperative Injection of Naldebain® in Management of Acute and Chronic Pain After Laparoscopic Bariatric Surgery
Brief Title: Naldebain for Pain Control After Bariatric Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Tu, Yuan-Kun, Professor of Orthopedics and Superintendent, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMRP-73109N
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Pain, Postoperative; Pain, Chronic; Bariatric Surgery; Obesity; Pharmacokinetics
Keywords: Nalbupine; Dinalbuphine sebacate; Naldebain; Opioid; Laparoscopic gastric sleeve surgery; Laparoscopic gastric bypass surgery
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Obesity | interventions — sebacoyl dinalbuphine ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Naldebain (active drug in solvent containing benzyl benzoate and sesame oil) or placebo drug (solvent containing benzyl benzoate and sesame oil) will be prepared by the clinical pharmacists in an identical injection syringe within 30 min before injection. The participants, anesthesiologists, surgeons, investigators and outcomes assessors will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naldebain group (Active Comparator): Patients assigned to Naldebain® group will receive a single intramuscular injection of dinalbuphine sebacate (150 mg in 2 ml solvent containing benzyl benzoate and sesame oil) into the gluteus muscles under ultrasound-guidance.
  Interventions: Drug: Dinalbuphine sebacate
- Placebo group (Placebo Comparator): Patients assigned to placebo group will receive a single intramuscular injection of 2 ml solvent containing benzyl benzoate and sesame oil into the gluteus muscles under ultrasound-guidance.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: Dinalbuphine sebacate — Naldebain dissolved in benzyl benzoate and sesame oil (a total volume of 2ml) will be prepared in a 5-ml syringe 30 min before administration. Intramuscular injection into the gluteal muscles will be performed by an anesthesiologist under sonography-guidance.
  Other Names: Naldebain ER®; Sebacoyl Dinalbuphine Ester Injection
  Arms: Naldebain group
Drug: Placebo solution — Benzyl benzoate and sesame oil served as placebo solution (a total volume of 2ml) will be prepared in a 5-ml syringe 30 min before administration. Intramuscular injection into the gluteal muscles will be performed by an anesthesiologist under sonography-guidance.
  Arms: Placebo group

SUMMARY:
Laparoscopic gastric sleeve and bypass surgeries the most common bariatric procedures for weight loss and improved management of metabolic syndromes. Patients may suffer from wound pain or referred pain after laparoscopic bariatric operation. Most importantly, 11.8% of these patients complained surgical-related pain one year after operation, and 8% of them required prolonged use of opioid to control chronic postoperative pain (CPSP). However, there are currently lack of clinical practice guidelines or recommendations for prevention of CPSP after laparoscopic abdominal surgery. Although regional block techniques (i.e. truncal block or intrathecal opioid) are considered as effective supplementary analgesic approaches to improve postoperative pain control, parenteral administration of analgesics remain as the mainstay for pain management of laparoscopic abdominal surgery. Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is an extended-release dinalbuphine sebacate, and is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. A number of clinical studies have shown that single-dose of pre-operative intramuscular administration of Naldebain® provides significantly higher analgesic effect up to 1 week in hemorrhoidectomy and laparotomy surgery with a well-tolerated safety profile. Therefore, this PI-initiated randomized, double-blind, placebo-control trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in patients receiving laparoscopic gastric sleeve or bypass surgery, and prevention of the development of CPSP after surgery. This study will also analyze the plasma levels of nalbuphine following a single intramuscular injection in obese patients.

DETAILED DESCRIPTION:
Clinical studies indicate that more than 80% of patients suffer from surgical-related pain in the first few days after major laparotomy or laparoscopic abdominal surgery and about 10% of these patients may develop chronic postoperative pain (CPSP), which can last up to several years after surgery. One of the major risk factors for developing CPSP is inadequate management of the acute postoperative pain. Laparoscopic gastric sleeve and bypass surgeries the most common bariatric procedures for weight loss and improved management of metabolic syndromes. Patients may suffer from wound pain or referred pain after laparoscopic bariatric operation. Most importantly, 11.8% of these patients complained surgical-related pain one year after operation, and 8% of them required prolonged use of opioid to control CPSP. However, there are currently lack of clinical practice guidelines or recommendations for prevention of CPSP after laparoscopic abdominal surgery. Although regional block techniques (i.e. truncal block or intrathecal opioid) are considered as effective supplementary analgesic approaches to improve postoperative pain control, parenteral administration of analgesics remain as the mainstay for pain management of laparoscopic abdominal surgery. Nalbuphine is a semi-synthetic opioid that acts as a mixed kappa opioid agonist and mu opioid antagonist, but its clinical applications in relieving acute postoperative pain is limited by the relatively short duration of action of 3-6h. Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is an extended-release dinalbuphine sebacate, and is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. A number of clinical studies have shown that single-dose of pre-operative intramuscular administration of Naldebain® provides significantly higher analgesic effect up to 1 week in hemorrhoidectomy and laparotomy surgery with a well-tolerated safety profile. Naldebain® has not been tested in laparoscopic bariatric surgery and its pharmacokinetic profiles in overweight patients are undetermined. Therefore, this PI-initiated randomized, double-blind, placebo-control trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in patients receiving laparoscopic gastric sleeve or bypass surgery, and prevention of the development of CPSP after surgery. This study will also analyze the plasma levels of nalbuphine following a single intramuscular injection in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to receive laparoscopic gastric sleeve surgery or laparoscopic gastric bypass surgery

Exclusion Criteria:

* Laparotomy bariatric surgery
* American Society of Anesthesiologists physical status > or =4
* Chronic opioid user
* Allergy to nalbuphine, benzyl benzoate or sesame oil
* Anticipated to receive ventilator support via an endotracheal tube after operation
* Not able for verbal pain assessment or not able to participate questionnaire survey

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain | 7 days after operation
  Pain score measured by visual analogue scale (VAS 1-10, a continuum scale in which 0 represents "no pain" and and 10 represents "worst pain.")
Total requirement dose of rescue analgesics | 7 days after operation
  Total doses of opioids, NSAIDs, COX-2 inhibitors administered

SECONDARY OUTCOMES:
Incidence of chronic post-surgical pain | 3 months after operation
  Pain that newly develops after operation and lasts >2 months and other causes of pain are excluded
Quality of life after surgery | 3 months after operation
  Quality of life will be assessed by the HRQoL SF -12 Questionnaire, which consists a physical component summary (PCS) and a mental component summary (MCS). The rating scales range from yes-no to likert scales, and the final score of PCS and MCS will be calculated by an algorithm (QualityMetric's SF-12v1®). Scores range from 0 to 100, in which lower scores mean lower health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Fuh Lam, MD, PhD, Principal Investigator — E-Da Hospital, Kaohsiung, Taiwan
Locations (1):
- E-Da Hospital, Yanchao, Kaohsiung, Taiwan